CLINICAL TRIAL: NCT00953355
Title: Effects of Metformin With or Without Folate Supplementation on Homocysteine Levels and Endothelium in Women With Polycystic Ovary Syndrome
Brief Title: Metformin and Folate Supplementation in Polycystic Ovary Syndrome (PCOS) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07/009
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2009-08

CONDITIONS: Polycystic Ovary Syndrome; Anovulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation | interventions — Folic Acid; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folate (Experimental): Folate plus metformin
  Interventions: Drug: Folate plus metformin
- Placebo (Placebo Comparator): Placebo plus metformin
  Interventions: Drug: Placebo plus metformin

INTERVENTIONS:
Drug: Folate plus metformin — A six-month course of metformin (1700 mg daily) plus folic acid (400 microgram daily).
  Arms: Folate
Drug: Placebo plus metformin — A six-month course of metformin (1700 mg daily) plus placebo
  Arms: Placebo

SUMMARY:
Context: Metformin administration in women with polycystic ovary syndrome (PCOS) improves hormonal and metabolic patterns with beneficial effects in terms of reproductive outcomes and intermediate cardiovascular disease risk factors. Furthermore, reduced folate and vitamin B12, and increased homocysteine (Hcy) levels have been found in type-2 diabetes mellitus patients treated with metformin.

Objective: To evaluate if metformin administration exerts any effects on Hcy levels, and if folate supplementation may improve endothelial structure and function in PCOS patients.

DETAILED DESCRIPTION:
Fifty patients affected by PCOS without additional metabolic or cardiovascular diseases grouped in two age- and body mass index-matched treatment arms.

Interventions: A six-month course of metformin (1700 mg daily) plus folic acid (400 microgram daily) (experimental group, n=25) or placebo (control group, n=25) supplementation.

In each patient were evaluated: Complete hormonal and metabolic patterns, serum Hcy, folate, vitamin B12, and endothelin-1 (ET-1) concentrations, brachial artery diameter at baseline (BAD-B) and after reactive hyperemia (BAD-RH), flow-mediated dilation (FMD), and intima-media thickness (IMT) on both common carotid arteries.

ELIGIBILITY:
Inclusion Criteria:

* PCOS

Exclusion Criteria:

* age <18 or >35 years
* BMI >35 kg/m2
* neoplastic, metabolic, hepatic, renal, and cardiovascular disorders
* Current or previous use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic and anti-obesity drugs or other hormonal drugs.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Endothelial structure and function | six months

SECONDARY OUTCOMES:
Clinical outcome Metabolic outcome Endocrine outcome | six months

CONTACTS AND LOCATIONS:
Locations (1):
- "Pugliese" Hospital, Catanzaro, Italy

REFERENCES:
- [Result] Palomba S, Falbo A, Giallauria F, Russo T, Tolino A, Zullo F, Colao A, Orio F. Effects of metformin with or without supplementation with folate on homocysteine levels and vascular endothelium of women with polycystic ovary syndrome. Diabetes Care. 2010 Feb;33(2):246-51. doi: 10.2337/dc09-1516. Epub 2009 Nov 23. PMID 19933994